CLINICAL TRIAL: NCT00436956
Title: A Phase II Study of AZD2171 in Metastatic Androgen Independent Prostate Cancer
Brief Title: AZD2171 to Treat Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Dahut Jr., M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070059; 07-C-0059
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: VEGF; Angiogenesis; Hormone-Refractory; Bone Metastases; Docetaxel-Resistant; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy; cediranib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD2171 in Prostate Cancer (Experimental): Cohort 1 (n=35) received 20 mg AZD2171 (Cediranib) orally daily. Cohort 2 (n=23) received prednisone 10 mg orally daily with 20 mg AZD2171.
  Interventions: Procedure: Magnetic Resonance Imaging (DCE-MRI); Drug: AZD2171; Drug: Prednisone

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging (DCE-MRI) — Scans evaluate tumor tissue and blood flow.
  Other Names: MRI
Drug: AZD2171 — 20 mg oral daily for 28 days
  Other Names: Cediranib
Drug: Prednisone — 10mg orally daily in combination with AZD2171 20mg daily.
  Other Names: Deltasone

SUMMARY:
Background:

* AZD2171 (Cediranib) is an experimental drug that inhibits formation of new blood vessels.
* Tumors need new blood vessels to grow. Preventing the growth of new blood vessels with AZD2171 may inhibit tumor growth.

Objectives:

-To determine the effectiveness and side effects of AZD2171 in patients with prostate cancer that has metastasized (spread beyond the primary site).

Eligibility:

* Males 18 years of age and older with androgen-independent prostate cancer that has metastasized.
* Patients must have received prior treatment with docetaxel.

Design:

Patients take one AZD2171 by mouth every day in 28-day treatment cycles and undergo the following procedures:

* 1- to 2-day hospitalization at the start of the study for biopsies and blood measurements to determine the level of AZD2171 in the bloodstream. Blood is drawn immediately before the first dose, and 0.25 hr, 0.5 hr, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 12 hr, 24 hr, and 48 hours after the dose is taken.
* Blood tests before starting treatment and then monthly to determine the level of vascular endothelial growth factor receptor ( VEGFR), a protein involved in blood vessel formation.
* Magnetic resonance imaging (MRI) scans once a month to evaluate blood flow.
* Tumor biopsies (optional) both before and after the second and sixth treatment cycles.
* Clinic visits every 4 weeks, including various routine and research blood tests, urine test and electrocardiogram.
* Computed tomography (CT) scan of the chest, abdomen, and pelvis every 8 weeks
* Bone scan every 8 weeks

Patients record all doses of AZD2171 taken or missed in a pill diary. They record their blood pressure at least once daily in a blood pressure diary.

Treatment may continue as long as the patient tolerates the AZD2171 and the cancer does not worsen.

...

DETAILED DESCRIPTION:
Background:

* AZD2171 (Cediranib) is an oral potent inhibitor of receptor tyrosine kinases which impact vascular endothelial growth factor-A (VEGF).
* VEGF appears important in blood vessel formation and disease progression in prostate cancer.
* No known effective therapy in patients with progressive androgen-independent prostate cancer after treatment with docetaxel.

Objectives:

* Primary objective of this study is to determine if AZD2171 is associated with a 30% 6 month probability of progression free survival in patients with metastatic androgen independent prostate cancer (AIPC) as determined by clinical and radiographic criteria.
* Secondary objective of this study will be demonstration of biologic effect by the drug in the patient and on the tumor (when possible). Correlative studies will be conducted on serially obtained tissue biopsies and white blood cell collections.
* Laboratory correlates will include elucidation of activation of components of the VEGFR2 and angiogenesis pathways and evaluation of endothelial cell adhesion molecules (released by damaged cells) using enzyme-linked immunosorbent assay (ELISA), pharmacogenetic analysis of kinase insert domain receptor (KDR) variants and single nucleotide polymorphisms, and pharmacokinetic characterization of AZD2171 activity.

Eligibility:

* Metastatic progressive androgen-independent prostate cancer.
* Prior treatment with docetaxel.
* May not have corrected QT interval (QTc ) greater than 470 msec or greater than 1+ proteinuria on 2 consecutive dipsticks no less than 1 week apart.

Design:

* Phase II trial with a two stage design. 12 patients enrolled in first cohort, if 2 or more are progression free at 6 months than enroll up to 35 evaluable patients. The ceiling will be set at 37 to allow for inevaluable patients.
* Starting dose 20 mg QD (every day) for all patients.
* Once two stage design is complete then prednisone 10 mg once per day will be given in combination with AZD2171. The total number of patients will be 23 for this portion of the protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have histopathological confirmation of prostate cancer by the Laboratory of Pathology of the National Cancer Institute (NCI), Pathology Department of the National Naval Medical Center or Pathology Department of Walter Reed Army Medical Center prior to entering this study. Patients whose pathology specimens are no longer available may be enrolled in the trial if the patient has a clinical course consistent with prostate cancer and available documentation from an outside pathology laboratory of the diagnosis. In cases where original tissue blocks or archival biopsy material is available, all efforts should be made to have the material forwarded to the research team for use in correlative studies.
  2. Patients must have metastatic progressive androgen-independent prostate cancer. There must be radiographic evidence of disease that has continued to progress despite hormonal agents. Progression requires that a measurable lesion is expanding, new lesions have appeared, and/or that prostatic specific antigen (PSA) is continuing to rise on successive measurements. Patients on flutamide must have disease progression at least 4 weeks after withdrawal. Patients on bicalutamide or nilutamide must have progression at least 6 weeks after withdrawal.
  3. Patients must have received prior therapy with docetaxel for androgen-independent prostate cancer. Any number of prior treatments are acceptable.
  4. Age greater than or equal to 18 years.
  5. Life expectancy of greater than 3 months.
  6. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
  7. Patients must have normal organ and marrow function as defined below:

     Absolute neutrophil count greater than or equal to 1,500/mcL

     Platelets greater than or equal to 100,000/mcL

     Hemoglobin greater than or equal to 8 g/dL

     Total bilirubin within normal institutional limits (unless with clinical Gilbert's syndrome)

     Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST(SGOT))/alanine aminotransferase/serum glutamic pyruvic transaminase (ALT(SGPT) less than or equal to 2.5 times institutional upper limit of normal

     Creatinine less than or equal to 1.5 times institutional upper normal institutional limits

     OR

     Creatinine clearance greater than 40 mL/min/1.3 m^2 for patients with creatinin levels above institutional normal as calculated by the Cockcroft Gault formula.
  8. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
  9. All patients who have not undergone bilateral surgical castration must continue suppression of testosterone production by appropriate usage of gonadotropin releasing hormone (GnRH) agonists or antagonists.
  10. Patients must not have other invasive malignancies (within the past three years with the exception of non-melanoma skin cancers or non-invasive bladder cancer).
  11. AZD2171 has been shown to terminate fetal development in the rat, as expected for a process dependent on VEGF signaling. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment.
  12. Ability to understand and the willingness to sign a written informed consent document.
  13. Patients must have a blood pressure of less than 140/90 at the time of enrollment. Details of antihypertensive treatment, if required, will be left up to the primary care physician.

EXCLUSION CRITERIA:

1. Patients who have had chemotherapy, radiotherapy, or major surgery within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
2. Patients may not be receiving any agents not approved by the Food and Drug Administration (FDA) within the past four weeks.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Mean QTc greater than 470 msec (with Bazett's correction) in screening electrocardiogram or history of familial long Q wave, T wave (QT) syndrome.
5. Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart.
6. Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2171.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-10-16 (Actual); Primary Completion 2010-02-01 (Actual); Study Completion 2014-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balbay MD, Pettaway CA, Kuniyasu H, Inoue K, Ramirez E, Li E, Fidler IJ, Dinney CP. Highly metastatic human prostate cancer growing within the prostate of athymic mice overexpresses vascular endothelial growth factor. Clin Cancer Res. 1999 Apr;5(4):783-9. PMID 10213213
- [Background] Beedassy A, Cardi G. Chemotherapy in advanced prostate cancer. Semin Oncol. 1999 Aug;26(4):428-38. PMID 10482185
- [Background] Belgore FM, Blann AD, Lip GY. Measurement of free and complexed soluble vascular endothelial growth factor receptor, Flt-1, in fluid samples: development and application of two new immunoassays. Clin Sci (Lond). 2001 May;100(5):567-75. PMID 11294698
- [Background] Huang J, Jochems C, Talaie T, Anderson A, Jales A, Tsang KY, Madan RA, Gulley JL, Schlom J. Elevated serum soluble CD40 ligand in cancer patients may play an immunosuppressive role. Blood. 2012 Oct 11;120(15):3030-8. doi: 10.1182/blood-2012-05-427799. Epub 2012 Aug 28. PMID 22932804
- [Result] Dahut WL, Madan RA, Karakunnel JJ, Adelberg D, Gulley JL, Turkbey IB, Chau CH, Spencer SD, Mulquin M, Wright J, Parnes HL, Steinberg SM, Choyke PL, Figg WD. Phase II clinical trial of cediranib in patients with metastatic castration-resistant prostate cancer. BJU Int. 2013 Jun;111(8):1269-80. doi: 10.1111/j.1464-410X.2012.11667.x. Epub 2013 Feb 18. PMID 23419134
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0059.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 20 mg AZD2171 Daily: Participants received 20 mg AZD2171 (Cediranib) orally daily.
- 20 mg AZD2171 + 10mg Prednisone Daily: Participants received 20 mg AZD2171 (Cediranib) orally daily plus 10mg prednisone.
Period: Overall Study
Arm/Group | 20 mg AZD2171 Daily | 20 mg AZD2171 + 10mg Prednisone Daily
Started | 36 | 23
Completed | 35 (One pt was not evaluable due to a cord compression on day 2 of therapy; was removed from the trial.) | 23
Not Completed | 1 | 0
Not completed — Not evaluable | 1 | 0

BASELINE CHARACTERISTICS:
Population: The cohorts are grouped together because the second cohort added prednisone to minimize toxicity/side effects.
Groups:
- All Participants - AZD2171 & Prednisone: This group combines participants who received 20 mg AZD2171 (Cediranib) orally daily (n=35), in addition to participants who received 20 mg AZD2171 (Cediranib) orally daily plus 10mg prednisone (n=23). One pt was not evaluable due to a cord compression on day 2 of therapy; was removed from the trial (n=1).
Arm/Group | All Participants - AZD2171 & Prednisone
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 39
Age, Continuous [Median (Full Range); unit: years] | 68.9 [51.4 to 79.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Afican-American | 3
  Asian | 1
  White | 52
  Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Participants With 6-month Progression-free Survival (PFS)
Description: PFS is the proportion of subjects who progress or die by 6 months after the start of the combined therapy. PFS is determined by prostatic specific antigen (PSA) consensus criteria and the Response Evaluation Criteria in Solid Tumors (RECIST). PSA consensus criteria is defined as PSA decline of >/= 50% or PSA progression. RECIST is defined as the following: Complete response (CR) is disappearance of all target lesions; partial response (PR) is at least a 30% decline in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; and stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease ((PD) at least a 20% increase in the sum of the LD of target lesions, or the appearance of one or more lesions), taking as reference the smallest sum LD since the treatment started. Data is estimated and the probability of PFS as a function of time was determined using the Kaplan-Meier method.
Time Frame: 6 months
Population: One participant was not evaluable owing to the development of a cord compression on day 2 of therapy and was subsequently removed from the trial. Since the prednisone was added to relieve toxicity & outcome data is based on response, the cohorts were analyzed together in terms of response. No suggestion prednisone significantly altered outcomes.
Measure: Number; unit: percent probability
Arm/Group | All Participants - AZD2171 & Prednisone
Number analyzed (Participants) | 58
percent probability | 43.9

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 61.5 months
Measure: Count of Participants; unit: Participants
Groups:
- All Participants- AZD2171 & Prednisone: This group combines participants who received 20 mg AZD2171 (Cediranib) orally daily (n=35), in addition to participants who received 20 mg AZD2171 (Cediranib) orally daily plus 10mg prednisone (n=23). One pt was not evaluable due to a cord compression on day 2 of therapy; was removed from the trial (n=1).
Arm/Group | All Participants- AZD2171 & Prednisone
Number analyzed (Participants) | 59
Participants | 59

3. Secondary Outcome: Number of Grade 2 Toxicities
Description: Here is the number of Grade 2 (moderate) toxicities.
Time Frame: 61.5 months
Population: Only 58 participants were evaluable for toxicity.
Measure: Number; unit: toxicities
Arm/Group | 20 mg AZD2171 Daily | 20 mg AZD2171 + 10mg Prednisone Daily
Number analyzed (Participants) | 35 | 23
toxicities
  Hypertension | 17 | 8
  Fatigue | 15 | 4
  Anorexia | 12 | 6
  Weight loss | 11 | 4
  Hypothyroidism | 7 | 6
  Dehydration | 8 | 2
  Prolonged QTc | 8 | 2
  Nausea | 7 | 3
  Diarrhea | 8 | 0
  Hypoalbuminemia | 5 | 3
  Proteinuria | 5 | 3
  Elevated alkaline phosphatase | 4 | 2
  Aspartate transaminase | 3 | 3
  Vomiting | 4 | 2
  Hyperbilirubinemia | 4 | 1
  Muscle weakness | 2 | 1

4. Secondary Outcome: Number of Grade 3 Toxicities
Description: Here is the number of Grade 3 (severe) toxicities.
Time Frame: 61.5 months
Population: Only 58 participants were evaluable for toxicity.
Measure: Number; unit: toxicities
Arm/Group | 20 mg AZD2171 Daily | 20 mg AZD2171 + 10mg Prednisone Daily
Number analyzed (Participants) | 35 | 23
toxicities
  Hypertension | 0 | 0
  Fatigue | 4 | 2
  Anorexia | 1 | 1
  Weight loss | 2 | 0
  Hypothyroidism | 0 | 0
  Dehydration | 3 | 3
  Prolonged QTc | 1 | 1
  Nausea | 1 | 0
  Diarrhea | 0 | 0
  Hypoalbuminemia | 0 | 0
  Proteinuria | 0 | 0
  Elevated alkaline phosphatase | 5 | 0
  Aspartate transaminase | 2 | 0
  Vomiting | 1 | 0
  Hyperbilirubinemia | 1 | 0
  Muscle weakness | 3 | 1

5. Secondary Outcome: Median Overall Survival
Description: Time from treatment start date until date of death or date last known alive.
Time Frame: 44 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 20 mg AZD2171 Daily | 20 mg AZD2171 + 10mg Prednisone Daily
Number analyzed (Participants) | 35 | 23
Months | 11.7 [6.8 to 15.0] | 9.9 [5.7 to 14.8]

6. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Time interval from start of treatment to documented evidence of disease progression.
Time Frame: up to 14.9 months based on a Kaplan-Meier analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 20 mg AZD2171 Daily | 20 mg AZD2171 + 10mg Prednisone Daily
Number analyzed (Participants) | 35 | 23
Months | 3.6 [2 to 14.9] | 3.7 [2 to 14.9]

7. Secondary Outcome: Response Per the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Response was evaluated by the RECIST. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease (PD)is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Every 2 cycles (approximately 56 days)
Population: One patient was not evaluable owing to the development of a cord compression on day 2 of therapy and was subsequently removed from the trial. Out of 59 patients, 39 had measurable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants - AZD2171 & Prednisone
Number analyzed (Participants) | 39
Participants
  Complete Response | 0
  Confirmed Partial Response | 6
  Unconfirmed Partial Response | 1
  Not Evaluable | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 61.5 months.
Arm/Group | All Participants - AZD2171 & Prednisone
All-Cause Mortality (participants affected / at risk) | 40/59
Serious Adverse Events (participants affected / at risk) | 59/59
Other Adverse Events (participants affected / at risk) | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants - AZD2171 & Prednisone (N=59)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 4 (6)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 5 (6)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 21 (28)
Anemia (Blood and lymphatic system disorders) | 15 (30)
Anorexia (Gastrointestinal disorders) | 21 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 12 (17)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Blood bilirubin increased (Metabolism and nutrition disorders) | 6 (6)
Blurred vision (Eye disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (13)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CPK increased (Metabolism and nutrition disorders) | 1 (1)
Cardiac disorders - Other, specify (Prolonged QTc) (Cardiac disorders) | 1 (1)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Confusion (Nervous system disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Creatinine increased (Metabolism and nutrition disorders) | 2 (2)
Death NOS (General disorders) | 40 (40)
Dehydration (Gastrointestinal disorders) | 18 (27)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (11)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Gastrointestinal disorders) | 3 (3)
Dysphasia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema limbs (Blood and lymphatic system disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 12 (15)
Eye disorders - Other, specify (CRAO) (Eye disorders) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 27 (37)
Fever (General disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (7)
Gum infection (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 26 (26)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (18)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7)
Hypotension (Vascular disorders) | 6 (9)
Hypothyroidism (Endocrine disorders) | 13 (13)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
INR increased (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations - Other, specify (Infection) (Infections and infestations) | 1 (2)
Intracranial hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Investigations - Other, specify (CPK) (Investigations) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Lymph gland infection (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 15 (25)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (16)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 6 (9)
Pleural effusion (Cardiac disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 8 (14)
Psychosis (Nervous system disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Rhinitis infective (Immune system disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 6 (6)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Venous injury (Vascular disorders) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (11)
Weight loss (General disorders) | 19 (24)
White blood cell decreased (Blood and lymphatic system disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants - AZD2171 & Prednisone (N=59)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Agitation (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 12 (15)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 6 (6)
Allergic rhinitis (Immune system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 7 (11)
Anorexia (Gastrointestinal disorders) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 15 (17)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Cervical lymh node) (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Metabolism and nutrition disorders) | 4 (4)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac disorders - Other, specify (Inverted T waves) (Cardiac disorders) | 1 (1)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Metabolism and nutrition disorders) | 5 (6)
Dehydration (Gastrointestinal disorders) | 1 (1)
Depression (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 35 (42)
Dizziness (Nervous system disorders) | 12 (13)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Ear and labyrinth disorders - Other, specify (Ear fullness) (Ear and labyrinth disorders) | 1 (1)
Edema face (Blood and lymphatic system disorders) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 8 (8)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Eye disorders - Other, specify (Opthalmoplegia/diplopia (double Vision)) (Eye disorders) | 1 (1)
Fatigue (General disorders) | 22 (25)
Fever (General disorders) | 2 (3)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Forced expiratory volume decreased (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (13)
Hematuria (Renal and urinary disorders) | 4 (4)
Hemoglobinuria (Metabolism and nutrition disorders) | 2 (2)
Hot flashes (Endocrine disorders) | 1 (1)
Hyperhidrosis (General disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 16 (19)
Infections and infestations - Other, specify (Upper resp) (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 3 (3)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (15)
Nervous system disorders - Other, specify (Staring spells) (Nervous system disorders) | 1 (1)
Oral hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 7 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Proteinuria (Metabolism and nutrition disorders) | 13 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal hemorrhage (Blood and lymphatic system disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Rhinorrhea) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Urinary frequency (Renal and urinary disorders) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Vomiting (Gastrointestinal disorders) | 11 (11)
Weight loss (General disorders) | 21 (22)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2010-05-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT00436956/Prot_000.pdf
  • Informed Consent Form (2009-12-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT00436956/ICF_001.pdf